CLINICAL TRIAL: NCT06697496
Title: Navigation and Artificial Intelligence Technology for Indigenous Virtual Education on Smoking Cessation (NAITIVE)
Brief Title: A Smartphone Application (QuitBot) for the Improvement of Smoking Cessation Among American Indians and Alaska Natives, NAITIVE Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RG1124884; NCI-2024-08892 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U19MD020533 (NIH); FHIRB0020651 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-04

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Interviews as Topic; Carbon Monoxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Random assignments will be concealed from participants and researchers throughout the trial. Follow-up data will be collected by survey research unit that will be blind to random assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (QuitBot chatbot) (Experimental): Participants participate in the QuitBot program which involves chatbot messages over 42 days. Therapy description withheld to protect the integrity of the study.
  Interventions: Device: QuitBot Smoking Cessation Chatbot Program; Other: Survey Administration; Other: Interview; Procedure: Carbon Monoxide Measurement
- Arm II (QuitBot texting) (Active Comparator): Participants participate in the QuitBot program which involves text messages over 42 days. Therapy description withheld to protect the integrity of the study.
  Interventions: Device: QuitBot Smoking Cessation Text Messaging Program; Other: Survey Administration; Procedure: Carbon Monoxide Measurement

INTERVENTIONS:
Device: QuitBot Smoking Cessation Chatbot Program — Participate in Quitbot chatbot program
  Other Names: QuitBot chatbot program
  Arms: Arm I (QuitBot chatbot)
Device: QuitBot Smoking Cessation Text Messaging Program — Participate in Quitbot texting program
  Other Names: QuitBot texting program
  Arms: Arm II (QuitBot texting)
Other: Survey Administration — Ancillary studies
Other: Interview — Ancillary studies
  Arms: Arm I (QuitBot chatbot)
Procedure: Carbon Monoxide Measurement — Ancillary studies
  Other Names: CMONOX

SUMMARY:
This clinical trial develops a chatbot smartphone application (app), QuitBot, and text messaging to help American Indians (AI) and Alaska Natives (AN) to quit smoking commercial tobacco (smoking cessation), and evaluates two remote smoking cessation programs to see how well they work for helping AI/AN people quit smoking commercial tobacco. AI/AN populations have one of the highest rates of commercial cigarette smoking of any racial and ethnic group in the United States (US). They also have a higher rate of developing smoking-related cancer but are less likely to quit smoking. The two programs are designed to provide personalized support in setting a smoking cessation goal, tasks to reach the smoking cessation goal, and motivation to remain smoke-free. This may help to keep participants engaged and support them in their quit efforts, and may improve smoking cessation among AI and AN.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms. Both groups receive access to a 42-day quit smoking program.

ARM I: Participants receive daily QuitBot program chatbot messages about the importance of quitting smoking, setting a quit date, preparing to quit, quitting, and maintaining abstinence over 42 days.

ARM II: Participants receive daily QuitBot text messages about the importance of quitting smoking, setting a quit date, preparing to quit, quitting, and maintaining abstinence over 42 days.

After completion of study intervention, participants are followed up at 3, 6, and 12 months and may be contacted thereafter for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying as American Indian or Alaska Native, either alone or in combination with other races
* Age 18 and older
* Smoking combustible cigarettes daily in the past year
* Interest in quitting smoking
* Interest in learning skills to quit smoking
* Willing to be randomly assigned
* Have daily access to their own Android or iPhone smartphone
* Ability to download a smartphone app
* Ability to read English
* Not currently (i.e., within past 30 days) using other smoking cessation interventions
* No prior participation in our studies
* No prior use of SFT
* No household or family member participating
* US residency for the next twelve months
* Willingness to complete follow-up assessments at the 3-, 6-, and 12-month follow-ups
* Providing email, phone number(s), and mailing address

Exclusion Criteria:

* The reverse of the inclusion criteria
* Pregnant or breastfeeding
* Use of other tobacco products (e.g., ceremonial use of tobacco, e-cigarettes) will be assessed but is not an exclusion criterion, as it would limit the study's generalizability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 772 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
30-day point prevalence abstinence (PPA) | At 12-months post-randomization
  Will use a logistic regression model and standard smoking cessation trial intent-to-treat analysis, with all missing outcomes will be coded as smoking. The model will adjust for stratification factors and baseline factors that are significantly related to the outcome. Sensitivity analyses will include: (1) multiple imputation of missing outcomes, (2) complete case analysis, and (3) carbon monoxide (CO)-verified results adjusted for use of other combustible nicotine-containing tobacco products at the 12-month follow-up-in order to differentiate them from use of cigarettes at 12 months.

SECONDARY OUTCOMES:
30-day PPA | At 3- and 6- months post-randomization
  Also 24-hour and 7-day PPA at the 3-, 6-, and 12- month follow-ups. Will use a logistic regression model and standard smoking cessation trial intent-to-treat analysis, with all missing outcomes will be coded as smoking. The model will adjust for stratification factors and baseline factors that are significantly related to the outcome. Sensitivity analyses will include: (1) multiple imputation of missing outcomes, (2) complete case analysis, and (3) CO-verified results adjusted for use of other combustible nicotine-containing tobacco products at the 12-month follow-up-in order to differentiate them from use of cigarettes at 12 months.
Measures of bond between user and conversational chatbot | At 3- and 6-months post-randomization
  Will be measured via four subscales of the 12-item Working Alliance Inventory for Tobacco (WAIT-12), with technology intervention adaptations similar to those of prior chatbot research. Will calculate the proportion of treatment effect explained by each of the mediators. Number of times participants engaged with the intervention will be adjusted in Poisson regressions that account for the number of prompts a participant received.
Agreement on goals of treatment | At 3- and 6-months post-randomization
  Will be measured via four subscales of the WAIT-12, with technology intervention adaptations similar to those of prior chatbot research. Will calculate the proportion of treatment effect explained by each of the mediators.
Agreement on tasks of treatment | At 3- and 6-months post-randomization
  Will be measured via four subscales of the WAIT-12, with technology intervention adaptations similar to those of prior chatbot research. Will calculate the proportion of treatment effect explained by each of the mediators.
User's sense that QuitBot understands their needs | At 3- and 6-months post-randomization
  Will be measured via four subscales of the WAIT-12, with technology intervention adaptations similar to those of prior chatbot research. Will calculate the proportion of treatment effect explained by each of the mediators.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The trial results data will be published on ClinicalTrials.gov. The de-identified scientific data will be made available as public use data to the research community in openICPSR. No PII or PHI data will be shared or available for secondary use.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified scientific data will be made available to other users no later than the time of publication of the primary outcomes, or at the end of the performance period, whichever comes first. The de-identified data deposited in openICPSR will be available to the research community in perpetuity.
Access Criteria: Members of the research community using this data must register with ICPSR and agree to the Terms of Use, which include limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, requiring immediate reporting of any disclosure of participant identity, and requiring users agree not to share or redistribute any data downloads.